CLINICAL TRIAL: NCT06022614
Title: Effect of Adding Dexmedetomidine As Adjuvant to Bupivacaine in Ultrasound Guided Erector Spinae Plane Block for Post Modified Radical Mastectomy Pain Management
Brief Title: Effect of Adding Dexmedetomidine As Adjuvant to Bupivacaine in US Guided ESPB for Post MRM Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abanoub Habib (Other)
Responsible Party: Sponsor-Investigator, Abanoub Habib, Dr, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: erector spinae plane block
Record Dates: First submitted 2023-08-04; First posted 2023-09-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Erector Spinae Plane Block
MeSH Terms: interventions — Bupivacaine; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients receiving Block with Bupivacaine only (Active Comparator): consists of patients receiving erector spinae plane block with Bupivacaine only
  Interventions: Drug: Use Bupivacaine 0.25% Injectable Solution
- Patients receiving Block using Bupivacaine with Dexmedetomidine (Active Comparator): consists of patients receiving erector spinae plane block using bupivacaine with Dexmedetomidine
  Interventions: Drug: Bupivacaine 0.25% Injectable Solution plus Dexmedetomidine

INTERVENTIONS:
Drug: Use Bupivacaine 0.25% Injectable Solution — Group A Patients receiving 20 ml Bupivacaine 0.25% added to 1 ml normal saline.
  Arms: Patients receiving Block with Bupivacaine only
Drug: Bupivacaine 0.25% Injectable Solution plus Dexmedetomidine — Group B Patients receiving 20 ml Bupivacaine 0.25% added to 1 ml dexmedetomidine
  Arms: Patients receiving Block using Bupivacaine with Dexmedetomidine

SUMMARY:
The aim of the study is to assess the effect of adding dexmedetomidine to bupivacaine in US guided erector spinae plane block in modified radical mastectomy surgeries , Using visual analogue score and post-operative narcotics consumption.

Peripheral nerve blocks are effective adjuvant options for pain management in breast surgeries. The use of Erector spinae plane block (ESPB) has been proven to be very effective in controlling pain and minimizing narcotic consumption after modified radical mastectomy surgeries.

Many adjuvants to local anaesthetics were used to improve the duration and intensity of the peripheral nerve block.

DETAILED DESCRIPTION:
Breast cancer is one of the most important medical problems in the female gender, since among every eight women, one will suffer from breast cancer during her lifetime.

Acute post-operative pain is very common after breast surgeries which requires adequate pain management. Different peripheral nerve blocks such as paravertebral block had been used as an analgesic option for breast surgeries.

Erector spinae plane block is a newer interfascial plane block first described in 2016 who used it for treating thoracic neuropathic pain by injecting a local anesthetic deep into the erector spinae muscle at the level of T5. Moreover, ESPB is a reasonable option, with clearly identifiable sonographic landmarks and LA needle insertion and injection locations.

Later studies have shown that ESPB can provide effective analgesia in breast surgeries.

ESPB is achieved by injecting the local anesthetics locally deep to erector spinae muscle surface, as a part of multimodal analgesia. Given that erector spinae muscles anatomically situate along the thoracolumbar spine, ESPB promotes an extensive craniocaudal spread.

Ultrasound is a non-invasive visualization technology that helps in capturing the anatomical structure of target tissues, it can help to guide the direction and depth of anesthesia puncture needles, thus reducing the risk of complications .

Adjuvants to local anesthetics, such as opioids, alpha 2 agonists, magnesium and dexamethasone may improve the duration and intensity of peripheral nerve blocks effect.

ELIGIBILITY:
Inclusion Criteria:

* Age:30-65years.
* Physical status: ASA I,II.
* BMI<35.
* Localized breast cancer

Exclusion Criteria:

* Age:<30 and >65 years.
* Refusal of procedure or participation in the study by the patient.
* Physical status: ASA III or above.
* History of allergy to the study drug.
* BMI>35.
* Bleeding disorders and coagulopathy.
* Psychiatric illness that may interfere with the study.
* Metastatic breast cancer.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-08-15 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
The primary outcome will be the first time to request rescue analgesia. | From the end of the surgery till 24 hours
  The investigators assess first time to request rescue analgesia according to A) pain score from 0 to 10 while 0 means no pain (best) and 10 means sever pain (worst).
The primary outcome will be the first time to request rescue analgesia | From the end of the surgery till 24 hours
  B) patient hemodynamics ex. Heart rate if patient is tachypneic (HR more than 100 beat/min) which is means that the patient is in pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Ain Shams University, Cairo, Egypt